CLINICAL TRIAL: NCT02008474
Title: Using a State-wide Initiative to Disseminate Effective Behavioral Weight Loss Strategies: Study 4
Brief Title: SHARE Study 4: Financial Incentives for Weight Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211699-14
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Online weight loss + Incentives for behavior 3 months (Active Comparator)
  Interventions: Behavioral: Online weight loss + incentives for behavior 3 months
- Online weight loss + Incentives for weight loss 3 months (Active Comparator)
  Interventions: Behavioral: Online weight loss + incentives for weight loss at month 3
- Online weight loss + Incentives for behavior 12 months (Active Comparator)
  Interventions: Behavioral: Online weight loss + Incentives for behavior 12 months
- Online weight loss + Incentives for weight loss 12 months (Active Comparator)
  Interventions: Behavioral: Online weight loss + Incentives for weight loss 12 months

INTERVENTIONS:
Behavioral: Online weight loss + incentives for behavior 3 months — Participants will receive monetary incentives for submitting their behavior change information into a study website
  Arms: Online weight loss + Incentives for behavior 3 months
Behavioral: Online weight loss + incentives for weight loss at month 3 — Participants will receive an incentive for meeting their weight loss goal at month 3.
  Arms: Online weight loss + Incentives for weight loss 3 months
Behavioral: Online weight loss + Incentives for behavior 12 months — Participants will receive incentives for submitting behavior change information over the course of 12 months.
  Arms: Online weight loss + Incentives for behavior 12 months
Behavioral: Online weight loss + Incentives for weight loss 12 months — Participants will be receive monetary incentives for reaching their weight loss goal at months 3 and 12.
  Arms: Online weight loss + Incentives for weight loss 12 months

SUMMARY:
The purpose of this study is to examine different types of monetary incentive paradigms for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI >=25kg/m2
* English speaking
* Age 18-70

Exclusion Criteria:

* Health problems that make weight loss or unsupervised exercise unsafe
* Current pregnancy or plan to become pregnant int he next 12 months
* Planned relocation
* Current participation in weight loss research study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
weight change from initial assessment to the 3-month follow-up assessment measured on a digital scale to the nearest 0.1-kilogram | 0 to 3 months

SECONDARY OUTCOMES:
weight change from the initial assessment to the 12 month assessment measured on a digital scale to the nearest 0.1-kilogram | 0 to 12 months
Weight change from the 3 month assessment to the 12 month assessment measured on a digital scale to the nearest 0.1-kilogram | 3 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rena Wing, PhD, Principal Investigator — The Miriam Hospital; Tricia M Leahey, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States